CLINICAL TRIAL: NCT04561284
Title: Carbohydrate-induced Resilience of the Gut Microbiome After Antibiotics Use
Acronym: CARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL73140.068.20 / METC20-025
Record Dates: First submitted 2020-09-08; First posted 2020-09-23 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Overweight and Obesity; Insulin Resistance; Dysbiosis
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Dysbiosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indigestible fiber supplementation (Experimental): Participants will receive an indigestible fiber supplementation (classified) for a period of 8 weeks. Thrice daily, they will take the fiber powder during their meals.
  Interventions: Dietary Supplement: Indigestible fiber (classified)
- Placebo supplementation (Placebo Comparator): Participants will receive placebo supplementation (Maltodextrin) for a period of 8 weeks. Thrice daily, they will take the fiber powder during their meals. The amount of maltodextrin taken will be isocaloric with the amount of indigestible fiber.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Indigestible fiber (classified) — Participants will be asked to ingest 12 grams of indigestible fiber powder per day for a period of 8 weeks. Three times daily, they will take 4 grams of powder with their meal.
  Arms: Indigestible fiber supplementation
Dietary Supplement: Placebo — Participants will be asked to ingest 6 grams of placebo powder per day for a period of 8 weeks. Three times daily, they will take 2 grams of powder with their meal.
  Arms: Placebo supplementation

SUMMARY:
The gut microbiome is a complex ecosystem with a wide range of functions, and it is thought that it can influence multiple processes in the human body. In turn, the composition and activity of the gut microbiome is affected by many factors as well.

Antibiotics can be very effective in treating bacterial infections, but they are also associated with detrimental health effects. Previous studies have already shown that antibiotics disturb the human gut microbiome composition by destroying commensal bacteria. As it is well known that the microbiome influences host metabolism, perturbation of the healthy microbiome (dysbiosis) is thought to be disease causing.

Prebiotics, on the other hand, are beneficial for the gut microbiome. These so-called indigestible fibers are naturally present in our foods, but cannot be metabolised by the human body. Many bacteria in the human gut are able to ferment these fibers and they subsequently produce beneficial products for the rest of the body. Besides this, fiber intake stimulates growth of commensal bacteria in the human gut.

Although it has become increasingly clear that prebiotics have a beneficial effect on the gut microbiome and general health, it is still unclear to which extent the beneficial effects of prebiotics supplementation occur after the gut microbiome is disturbed by antibiotics. We hypothesize that prebiotic supplementation after antibiotics use will improve restoration of the gut microbiome to a healthy state compared to placebo.

DETAILED DESCRIPTION:
In this double-blind, randomized placebo-controlled study, 40 overweight, but otherwise healthy adults will first receive vancomycin for 7 days (3x 500mg per day) to disturb the gut microbiome. They will then receive either indigestible fiber supplementation (classified) ór a placebo for the following 8 weeks. All study parameters will be assessed in two parallel groups, to which subjects will be assigned using minimization.

After initial screening, participants will be asked to visit the university for a total of 6 times during a period of 11 weeks. A clinical investigation day will take place at baseline, after antibiotics use and after the supplementation period. The remaining 3 visits will be short visits during the supplementation period (week 2, 4 & 6 of supplementation). Participants will be asked to collect feces every day before the university visits.

During the clinical investigation days, an abdominal subcutaneous adipose tissue will be taken under fasting conditions. Participants will also perform a 7-point oral glucose tolerance test to assess their insulin sensitivity. Furthermore, blood samples will be taken in the fasted state to assess markers of fat metabolism, short-chain fatty acids, gut hormones and inflammatory markers. Participants will be asked to hand in collected feces and to fill in questionnaires regarding stool consistency, stool frequency and physical activity. Lastly, they will be asked to hand in filled-in 3-day food diaries.

On the 3 remaining visits during the supplementation period, participants will hand in collected feces and food diaries, and fill in the questionnaires.

For these 6 visits, participants will have to invest approximately 14 hours.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (BMI: 25 - 35 kg/m^2)
* Caucasian
* Stable body weight (< 3 kg change) for the last 3 months

Exclusion Criteria:

* Known allergic reaction to vancomycin or other glycopeptide antibiotics;
* Pre-diabetes, diabetes mellitus, cardiovascular disease, kidney disease, hearing disorders, cancer, asthma or bronchitis, liver malfunction, diseases affecting glucose tolerance, major illness with a life expectancy < 5 years, gastrointestinal disease or abdominal surgery;
* Abuse of products; alcohol and drugs, excessive nicotine use (> 20 cigarettes per day);
* Regular use of laxation products;
* Use of antibiotics in the past 3 months;
* Regular supplementation of pre- or probiotic products, use of pre- or probiotics 3 months prior to the start of the study;
* Plans to lose weight or currently following a hypocaloric diet;
* Following a vegetarian diet;
* Participation in organized sports activities for > 3 hours per week;
* Suffering from hearing loss or other hearing problems;
* Currently pregnant, planning to become pregnant, or currently breastfeeding.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition | Change in gut microbiota composition after antibiotic use (week 1) compared to baseline & change in microbial composition during fiber supplementation (week 3, 5, 7 & 9) compared to placebo.
  Fecal samples will be collected at baseline, week 1, 3, 5, 7 and 9. Microbial DNA will be extracted, and microbiota composition will be analyzed by next-generation sequencing.
  Gut microbiota composition at week 1 will be compared with baseline to assess the effect of antibiotic use. Microbial composition during the supplementation period (week 3, 5, 7 & 9) will be compared between the two study arms to assess restorative potential of the indigestible fiber.
Gut microbiota activity | Change in gut microbiota activity after antibiotic use (week 1) compared to baseline & change in microbial activity during fiber supplementation (week 3, 5, 7 & 9) compared to placebo.
  Fecal samples will be collected at baseline, week 1, 3, 5, 7 and 9. Microbial proteins will be analyzed by mass spectrometry (MS) after extraction.
  Gut microbiota activity at week 1 will be compared with baseline to assess the effect of antibiotic use. Microbial activity during the supplementation period (week 3, 5, 7 & 9) will be compared between the two study arms to assess restorative potential of the indigestible fiber.
Fecal Short-Chain Fatty Acids (SCFA) | Change in fecal SCFA levels after antibiotic use (week 1) compared to baseline & change in fecal SCFA levels during fiber supplementation (week 3, 5, 7 & 9) compared to placebo.
  Fecal samples will be collected at baseline, week 1, 3, 5, 7 and 9. Fecal SCFA levels will be analyzed using gas-chromatography MS.
  Fecal SCFA levels at week 1 will be compared with baseline levels to assess the effect of antibiotic use. SCFA levels in feces during the supplementation period (week 3, 5, 7 & 9) will be compared between the two study arms to assess restorative potential of the indigestible fiber.
Resistome analysis | Change in ARG presence after antibiotic use (week 1) compared to baseline & change in ARG presence during fiber supplementation (week 3, 5, 7 & 9) compared to placebo.
  Fecal samples will be collected at baseline, week 1, 3, 5, 7 and 9. Microbial DNA will be extracted, and resistome analysis will be performed via qPCR, targeting specific antibiotic resistance genes (ARG).
  Presence of ARG at week 1 will be compared with baseline to assess the effect of antibiotic use. ARG presence during the supplementation period (week 3, 5, 7 & 9) will be compared between the two study arms to assess the effect of the indigestible fiber.

SECONDARY OUTCOMES:
Body Mass Index | Change in BMI after 1 week of antibiotic use compared to baseline & after 8-week indigestible fiber supplementation compared to placebo.
  At the clinical investigation days (baseline, week 1 and week 9), Body Mass Index will be measured.
Insulin sensitivity | Change in insulin sensitivity after 1 week of antibiotic use compared to baseline & after 8-week indigestible fiber supplementation compared to placebo.
  At the 3 clinical investigation days, a 7-point oral glucose tolerance test will be performed to assess insulin sensitivity. Glucose and insulin levels in the blood will be measured, and HOMA-IR will be calculated.
Plasma markers of fat metabolism | Change in markers of fat metabolism after 1 week of antibiotic use compared to baseline & after 8-week indigestible fiber supplementation compared to placebo.
  At the 3 clinical investigation days, blood will be drawn in the fasted state to analyze plasma Free Fatty Acid and Triacylglycerol levels.
Adipose tissue gene expression | Change in adipose tissue gene expression after 1 week of antibiotic use compared to baseline & after 8-week indigestible fiber supplementation compared to placebo.
  At the 3 clinical investigation days, an abdominal subcutaneous adipose tissue biopsy will be taken to investigate adipose tissue gene expression. Expression of genes of interest will be analysed using targeted qPCR.
Adipose tissue protein levels | Change in adipose tissue protein levels after 1 week of antibiotic use compared to baseline & after 8-week indigestible fiber supplementation compared to placebo.
  At the 3 clinical investigation days, an abdominal subcutaneous adipose tissue biopsy will be taken to investigate adipose tissue protein levels. Proteins of interest will be analysed using Western Blot.
Plasma short chain fatty acids | Change in plasma SCFA levels after 1 week of antibiotic use compared to baseline & after 8-week indigestible fiber supplementation compared to placebo.
  At the 3 clinical investigation days, blood will be drawn in the fasted state to analyse levels of the SCFA acetate, butyrate and propionate.
Inflammatory markers | Change in plasma inflammatory marker levels after 1 week of antibiotic use compared to baseline & after 8-week indigestible fiber supplementation compared to placebo.
  At the 3 clinical investigation days, blood will be drawn in the fasted state to analyse levels of the inflammatory markers IL-6, IL-8, MCP1, TNF-alpha, leptin, adiponectin and LBP.
Gut hormones | Change in plasma gut hormone levels after 1 week of antibiotic use compared to baseline & after 8-week indigestible fiber supplementation compared to placebo.
  At the 3 clinical investigation days, blood will be drawn in the fasted state to analyse levels of the gut hormones GLP-1 and PYY.

OTHER OUTCOMES:
Dietary intake | Comparing dietary intake at week 1, 3, 5, 7 & 9 with baseline.
  Participants will be asked to fill in a three-day food diary. These will be used to check dietary intake during the weight management period, versus baseline. This will also serve as a measure of compliance with dietary advice.
Physical activity | Comparing physical activity at week 1, 3, 5, 7 & 9 with baseline.
  At all 6 visits, participants will be asked to fill in the SQUASH-questionnaire for physical activity. These will be used to check physical activity.
Stool consistency | Comparing stool consistency at week 1, 3, 5, 7 & 9 with baseline.
  Participants will be asked to fill in the Bristol Stool Chart on the day prior to each of the 6 visits, in order assess stool consistency.
Gastrointestinal symptoms | Comparing gastrointestinal symptoms at week 1, 3, 5, 7 & 9 with baseline.
  Participants will be asked to fill in the Gastrointestinal Symptom Rating Scale on the day prior to each of the 6 visits, in order to assess potential gastrointestinal complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, Prof. Dr., Principal Investigator — Department of Human Biology, Maastricht University
Locations (1):
- Department of Human Biology, Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No